CLINICAL TRIAL: NCT04454840
Title: A Clinical Study on Safety and Effectiveness of Intravenous Infusion Plasma From Healthy Young People to Treat Amyotrophic Lateral Sclerosis
Brief Title: Treatment of Intravenous Infusion Plasma in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUTH2017118
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Plasma infusion
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Riluzole

STUDY DESIGN:
Masking Description: Open Lable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological+Riluzole (Experimental): Plasma from healthy young people treatment + Riluzole
  Interventions: Biological: Plasma from healthy young people treatment + Riluzole
- Riluzole (Active Comparator): Riluzole
  Interventions: Drug: Riluzole

INTERVENTIONS:
Biological: Plasma from healthy young people treatment + Riluzole — Intravenous injection: the subjects received 400ml of intravenous plasma infusion every 2 weeks, with a continuous course of 2 treatments and a course of treatment every 3 months. The course of treatment lasted 10 months, with a total of 3200ml of plasma infusion.
  Arms: Biological+Riluzole
Drug: Riluzole — The basic treatment is Riluzole 25~50mg twice daily
  Arms: Riluzole

SUMMARY:
To evaluate the safety and effectiveness of intravenous infusion of plasma from healthy young people for the treatment of amyotrophic lateral sclerosis.

DETAILED DESCRIPTION:
This is a single-center, open-label clinical study to evaluate the safety and effectiveness of intravenous infusion of plasma from healthy young people for the treatment of amyotrophic lateral sclerosis. The main outcome indicators are the record of adverse reactions and the rate of change of amyotrophic lateral sclerosisFunctional Rating Scale score. The secondary outcome indicators include survival time-time to the end event (death, tracheotomy, continuous ventilator dependence), forced vital capacity (FVC), recognition Knowledge function evaluation (ECAS score).

ELIGIBILITY:
Inclusion Criteria:

* Meet the following diagnosis standard: confirmed, proposed and laboratory supported diagnosis;
* Age 50-70 years old ;
* 3-18 months course of disease;
* Forced vital capacity (FVC) ≥70% predicted value;
* Total amyotrophic lateral sclerosis Functional Rating Scale score ≥36, scores of respiratory related items ≥10;
* Take Riluzole regularly before participate in this trial (25~50mg twice a day for at least 30 days continuously) without obvious side effects and can continue to take for 22 months;
* Participants of childbearing age take reasonable and effective contraceptive measures from the time of enrollment to the end of follow-up;
* Signed informed consent.

Exclusion Criteria:

* Familial amyotrophic lateral sclerosis;
* Female during pregnancy and lactation;
* Positive hepatitis B, hepatitis C or HIV in screening
* History of cytomegalovirus and malaria infection;
* After tracheotomy and ventilator-dependent state (daily use of non-invasive ventilator ≥ 22 hours for 7 consecutive days);
* After percutaneous gastrostomy (PEG) operation;
* Has had allergic reactions and other adverse reactions during blood transfusion;
* Have diseases of the blood system (including Immunoglobulin A deficiency);
* alanine transaminase, Aspartate transaminase≥ 3 times the upper limit of normal;
* Abnormal renal function (Cr, BUN);
* History of malignant tumors;
* Combining severe cardiopulmonary diseases, autoimmune diseases, mental diseases, substance abuse history, etc;
* Currently participating in other clinical studies or using other drugs in researching.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Amyotrophic lateral sclerosis Functional Rating Scale scores | 22 months after intervention
  Rate of amyotrophic lateral sclerosis Functional Rating Scale scores changes

SECONDARY OUTCOMES:
Survival time | 22 months after intervention
  The time of the end event (death, tracheotomy, continuous ventilator dependence);
Forced vital capacity (FVC) | 22 months after intervention
  The change from baseline to the end of follow-up;
Cognitive function evaluation (ECAS score) | 22 months after intervention
  The change from baseline to the end of follow-up;

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No